CLINICAL TRIAL: NCT04344704
Title: Prevention of Inappropriate Therapies and Serious Adverse Cardiac and Cerebrovascular Events With a Single Chamber Implantable Cardioverter Defibrillator (ICD) With DX Floating Dipole Detection. PREVENT DX
Brief Title: Prevention of Inappropriate Therapies and MACCE With a Single Chamber ICD With DX Floating Dipole Atrial Detection
Acronym: PREVENT-DX
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Trialance SCCL (Industry)
Responsible Party: Sponsor
Other Study IDs: DX01
Record Dates: First submitted 2020-04-02; First posted 2020-04-14 (Actual); Last update posted 2020-04-14 (Actual); Status verified 2020-04

CONDITIONS: Prevention of Inappropriate Therapies and MACCE. Single-chamber ICD

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- DX devices with SMART headset detection enabled: The SMART detection algorithm is designed to, with the aid of atrial rhythm assessment, discriminate between ventricular tachycardias and a variety of supraventricular tachyarrhythmias for which device intervention is not required or desired
  Interventions: Other: Single chamber DAI device with floating atrial dipole
- DX device programmed in single chamber mode: with the activation of one of the available discrimination criteria:
  * Onset: distinguishes slow onset or onset tachycardias from sudden onset
  * Stability: distinguishes between irregularly transmitted supraventricular tachycardias and ventricular tachycardias requiring therapy by continuous interval monitoring.
  * Morphmatch: helps to distinguish between supra and ventricular signals through analysis of episode QRS width
  Interventions: Other: Single chamber DAI device with floating atrial dipole

INTERVENTIONS:
Other: Single chamber DAI device with floating atrial dipole — DAI for the detection of atrial signals with optimized programming, using Smart, Onset & Stability, and Morphmatch methods

SUMMARY:
Prevention of inappropriate therapies and serious adverse cardiac and cerebrovascular events with a single chamber implantable defibrillator with DX floating dipole atrial detection

DETAILED DESCRIPTION:
Prospective, randomized, open-label, multicenter, international study in a population with an accepted indication for an implantable automatic defibrillator.

The main objective is to know the different values of the rates of inappropriate therapies, of serious cardiac and cerebrovascular adverse events, and of the appropriate detections in single-chamber ICD devices, with optimized programming according to the patient's arrhythmic history, using the three discrimination methods. arrhythmias: Smart, Onset and Stability, and Morphmatch.

The device under investigation is a single chamber with a floating atrial dipole for the detection of atrial signals.

Patients who are included in the study will present an indication for an automatic cardioverter-defibrillator device according to clinical practice guidelines for an ICD and who also do not have an indication for permanent stimulation in the right atrium. For this reason, the indication of patients will be those that require an ICD without the implantation of an electrode in the atrium, that is, single-chamber ICDs or DX ICDs since both, from the therapeutic point of view, are equivalent.

The centers will follow standard clinical practice to diagnose patients

ELIGIBILITY:
Inclusion Criteria:

* Patients with an indication of a single chamber ICD due to high risk of sudden death.
* Patients with and without a prior history of AF.
* Patients with indication for primary and secondary prevention.
* Device optimized for the discrimination of supraventricular events.
* DX device implant with single floating cable.
* Activation of "Home Monitoring" function.
* Over 18 years.
* Signature of informed consent

Exclusion Criteria:

* Indication for permanent atrial pacing according to current pacing guidelines.
* Congestive heart failure grade IV.
* Candidates for Cardiac Resynchronization Therapy.
* Patients with a previous device.
* Permanent Atrial Fibrillation.
* Life expectancy less than 12 months.
* Pregnant or lactating women.
* Patients who are unable to understand the nature of the study.
* Subjects with irreversible brain damage caused by pre-existing brain disease.
* Heart transplant 6 months prior to recruitment or expected in the next 3 months.
* Cardiac surgery 3 months prior to recruitment or planned for the next 3 months.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Population with an accepted indication for an implantable automatic defibrillator
Sampling Method: Probability Sample
Enrollment: 462 (Estimated)
Dates: Start 2018-11-02 (Actual); Primary Completion 2022-09 (Estimated); Study Completion 2023-03 (Estimated)

PRIMARY OUTCOMES:
The combined rate of inappropriate therapies and serious adverse cardiac and cerebrovascular events (MACCE) single-chamber devices with floating atrial dipole with the Smart function activated | 24 months
  determine the combined rate is not less than in single-chamber devices without atrial detection using any of the supraventricular arrhythmia discrimination modalities: Onset and Stability, and Morphmatch.

SECONDARY OUTCOMES:
Inappropriate therapies distribution | 24 months
  According to the type of indication for an ICD in primary and secondary prevention
Programming adjustment justification | 24 months
  Adjustments suggested by the European Heart Rhythm Association
Distribution of inappropriate therapies by chosen schedule | 24 months
Proportion of appropriate and inappropriate diagnoses | 24 months
  By diagnosis group
Differences in events according to Onset & Stability method versus Morphmatch method | 24 months
  Events in single chamber programming without floating dipole
Appropriate therapies by group and by indication | 24 months
  Portion of appropriate therapies
Triggers of Inappropriate therapies | 24 months
Patients presenting atrial fibrillation before inclusion | 24 months
  percentage
Patients with no prior history of atrial fibrillation (AF) who have AF during study follow-up | 24 months
  Percentage
General atrial load in patients with and without previous manifestation of atrial fibrillation | 24 months
Percentage of patients with clinical AF (atrial fibrillation) versus subclinical AF (<6 minutes duration). | 24 months
  Clinical AF meaning > 6 minutes duration and subclinical AF meaning <6 minutes duration
Cerebrovascular events presenting previous episodes of atrial fibrillation | 24 months
  Rate

CONTACTS AND LOCATIONS:
Overall Officials: Ignacio Fernández Lozano, MD, Principal Investigator — Hospital Universitario Puerta de Hierro (HUPH)
Locations (16):
- Spain (16):
  - Hospital Universitario Clínico de Santiago, Santiago de Compostela, A Coruña
  - Hospital Universitario de Araba, Vitoria-Gasteiz, Alava
  - Hospital Universitario Germans Trias i Pujol, Badalona, Barcelona
  - Hospital Universitario de Bellvitge, L'Hospitalet de Llobregat, Barcelona
  - Hospital Universitario de Donostia, Donostia / San Sebastian, Guipúzcoa
  - Hospital Universitario Puerta de Hierro, Majadahonda, Madrid
  - Hospital Álvaro Cunqueiro, Vigo, Pontevedra
  - Complejo Hospitalario Universitario de Canarias, Santa Cruz de Tenerife, Tenerife
  - Complejo Hospitalario Universitario A Coruña, A Coruña
  - Hospital Universitario Josep Trueta, Girona
  - Hospital San Pedro, Logroño
  - Hospital Universitario La Paz, Madrid
  - Hospital Universitario Virgen de la Victoria, Málaga
  - Hospital Universitario de Tarragona Joan XXIII, Tarragona
  - Hospital Universitario y Politécnico La Fe, Valencia
  - Hospital Clínico y Universitario de Valladolid, Valladolid

REFERENCES:
- [Result] Guedon-Moreau L, Kouakam C, Klug D, Marquie C, Brigadeau F, Boule S, Blangy H, Lacroix D, Clementy J, Sadoul N, Kacet S. Decreased delivery of inappropriate shocks achieved by remote monitoring of ICD: a substudy of the ECOST trial. J Cardiovasc Electrophysiol. 2014 Jul;25(7):763-70. doi: 10.1111/jce.12405. Epub 2014 Apr 10. PMID 24602062
- [Result] Kolb C, Sturmer M, Sick P, Reif S, Davy JM, Molon G, Schwab JO, Mantovani G, Dan D, Lennerz C, Borri-Brunetto A, Babuty D. Reduced risk for inappropriate implantable cardioverter-defibrillator shocks with dual-chamber therapy compared with single-chamber therapy: results of the randomized OPTION study. JACC Heart Fail. 2014 Dec;2(6):611-9. doi: 10.1016/j.jchf.2014.05.015. Epub 2014 Oct 1. PMID 25282033
- [Result] Boles U, Gul EE, Fitzgerald L, Sadiq Ali F, Nolan C, Aldworth-Gaumond K, Redfearn DR, Baranchuk A, Glover B, Simpson C, Abdollah H, Michael KA. Standardized programming to reduce the burden of inappropriate therapies in implantable cardioverter defibrillators - Single centre follow up results. Indian Pacing Electrophysiol J. 2018 Mar-Apr;18(2):56-60. doi: 10.1016/j.ipej.2017.10.010. Epub 2017 Oct 27. PMID 29111168
- [Result] van Rees JB, Borleffs CJ, de Bie MK, Stijnen T, van Erven L, Bax JJ, Schalij MJ. Inappropriate implantable cardioverter-defibrillator shocks: incidence, predictors, and impact on mortality. J Am Coll Cardiol. 2011 Feb 1;57(5):556-62. doi: 10.1016/j.jacc.2010.06.059. PMID 21272746
- [Result] Moss AJ, Schuger C, Beck CA, Brown MW, Cannom DS, Daubert JP, Estes NA 3rd, Greenberg H, Hall WJ, Huang DT, Kautzner J, Klein H, McNitt S, Olshansky B, Shoda M, Wilber D, Zareba W; MADIT-RIT Trial Investigators. Reduction in inappropriate therapy and mortality through ICD programming. N Engl J Med. 2012 Dec 13;367(24):2275-83. doi: 10.1056/NEJMoa1211107. Epub 2012 Nov 6. PMID 23131066
- [Result] Kutyifa V, Moss AJ, Schuger C, McNitt S, Polonsky B, Ruwald AH, Ruwald MH, Daubert JP, Zareba W. Reduction in Inappropriate ICD Therapy in MADIT-RIT Patients Without History of Atrial Tachyarrhythmia. J Cardiovasc Electrophysiol. 2015 Aug;26(8):879-884. doi: 10.1111/jce.12692. Epub 2015 Jun 15. PMID 25917337
- [Result] Vanhees L, Kornaat M, Defoor J, Aufdemkampe G, Schepers D, Stevens A, Van Exel H, Van Den Beld J, Heidbuchel H, Fagard R. Effect of exercise training in patients with an implantable cardioverter defibrillator. Eur Heart J. 2004 Jul;25(13):1120-6. doi: 10.1016/j.ehj.2004.04.034. PMID 15231370
- [Result] Sterns LD, Meine M, Kurita T, Meijer A, Auricchio A, Ando K, Leng CT, Okumura K, Sapp JL, Brown ML, Lexcen DR, Gerritse B, Schloss EJ. Extended detection time to reduce shocks is safe in secondary prevention patients: The secondary prevention substudy of PainFree SST. Heart Rhythm. 2016 Jul;13(7):1489-96. doi: 10.1016/j.hrthm.2016.03.022. Epub 2016 Mar 14. PMID 26988379
- [Result] Auricchio A, Hudnall JH, Schloss EJ, Sterns LD, Kurita T, Meijer A, Fagan DH, Rogers T. Inappropriate shocks in single-chamber and subcutaneous implantable cardioverter-defibrillators: a systematic review and meta-analysis. Europace. 2017 Dec 1;19(12):1973-1980. doi: 10.1093/europace/euw415. PMID 28340005
- [Result] Boersma L, Barr C, Knops R, Theuns D, Eckardt L, Neuzil P, Scholten M, Hood M, Kuschyk J, Jones P, Duffy E, Husby M, Stein K, Lambiase PD; EFFORTLESS Investigator Group. Implant and Midterm Outcomes of the Subcutaneous Implantable Cardioverter-Defibrillator Registry: The EFFORTLESS Study. J Am Coll Cardiol. 2017 Aug 15;70(7):830-841. doi: 10.1016/j.jacc.2017.06.040. PMID 28797351
- [Result] Cay S, Canpolat U, Ucar F, Ozeke O, Ozcan F, Topaloglu S, Aras D. Programming implantable cardioverter-defibrillator therapy zones to high ranges to prevent delivery of inappropriate device therapies in patients with primary prevention: results from the RISSY-ICD (Reduction of Inappropriate ShockS bY InCreaseD zones) trial. Am J Cardiol. 2015 May 1;115(9):1235-43. doi: 10.1016/j.amjcard.2015.01.558. Epub 2015 Feb 12. PMID 25765588
- [Result] Defaye P, Boveda S, Klug D, Beganton F, Piot O, Narayanan K, Perier MC, Gras D, Fauchier L, Bordachar P, Algalarrondo V, Babuty D, Deharo JC, Leclercq C, Marijon E, Sadoul N; DAI-PP Investigators. Dual- vs. single-chamber defibrillators for primary prevention of sudden cardiac death: long-term follow-up of the Defibrillateur Automatique Implantable-Prevention Primaire registry. Europace. 2017 Sep 1;19(9):1478-1484. doi: 10.1093/europace/euw230. PMID 28340096
- [Result] Kreuz J, Balta O, Liliegren N, Mellert F, Esmailzadeh B, Nickenig G, Schwab JO. Incidence and characteristics of appropriate and inappropriate therapies in recipients of ICD implanted for primary prevention of sudden cardiac death. Pacing Clin Electrophysiol. 2007 Jan;30 Suppl 1:S125-7. doi: 10.1111/j.1540-8159.2007.00621.x. PMID 17302687
- [Result] Konstantino Y, Haim M, Boxer J, Goldenberg I, Feldman A, Michowitz Y, Glikson M, Suleiman M; Israeli Working Group on Pacing and Electrophysiology. Clinical Outcomes of Single- versus Dual-Chamber Implantable Cardioverter Defibrillators: Lessons from the Israeli ICD Registry. J Cardiovasc Electrophysiol. 2016 Jun;27(6):718-23. doi: 10.1111/jce.12953. Epub 2016 Mar 18. PMID 26852908
- [Result] Oginosawa Y, Kohno R, Honda T, Kikuchi K, Nozoe M, Uchida T, Minamiguchi H, Sonoda K, Ogawa M, Ideguchi T, Kizaki Y, Nakamura T, Oba K, Higa S, Yoshida K, Tsunoda S, Fujino Y, Abe H. Superior Rhythm Discrimination With the SmartShock Technology Algorithm - Results of the Implantable Defibrillator With Enhanced Features and Settings for Reduction of Inaccurate Detection (DEFENSE) Trial. Circ J. 2017 Aug 25;81(9):1272-1277. doi: 10.1253/circj.CJ-16-1330. Epub 2017 Apr 20. PMID 28428489
- [Result] Schwab JO, Bonnemeier H, Kleemann T, Brachmann J, Fischer S, Birkenhauer F, Eberhardt F. Reduction of inappropriate ICD therapies in patients with primary prevention of sudden cardiac death: DECREASE study. Clin Res Cardiol. 2015 Dec;104(12):1021-32. doi: 10.1007/s00392-015-0870-z. Epub 2015 May 23. PMID 26002818
- [Result] Kloppe A, Proclemer A, Arenal A, Lunati M, Martinez Ferrer JB, Hersi A, Gulaj M, Wijffels MC, Santi E, Manotta L, Mangoni L, Gasparini M. Efficacy of long detection interval implantable cardioverter-defibrillator settings in secondary prevention population: data from the Avoid Delivering Therapies for Nonsustained Arrhythmias in ICD Patients III (ADVANCE III) trial. Circulation. 2014 Jul 22;130(4):308-14. doi: 10.1161/CIRCULATIONAHA.114.009468. Epub 2014 May 16. PMID 24838360
- [Result] Friedman PA, Bradley D, Koestler C, Slusser J, Hodge D, Bailey K, Kusumoto F, Munger TM, Militanu A, Glikson M. A prospective randomized trial of single- or dual-chamber implantable cardioverter-defibrillators to minimize inappropriate shock risk in primary sudden cardiac death prevention. Europace. 2014 Oct;16(10):1460-8. doi: 10.1093/europace/euu022. Epub 2014 Jun 13. PMID 24928948
- [Result] Worden NE, Alqasrawi M, Krothapalli SM, Mazur A. "Two for the Price of One": A Single-Lead Implantable Cardioverter-Defibrillator System with a Floating Atrial Dipole. J Atr Fibrillation. 2016 Apr 30;8(6):1396. doi: 10.4022/jafib.1396. eCollection 2016 Apr-May. PMID 27909501
- [Result] Wilkoff BL, Fauchier L, Stiles MK, Morillo CA, Al-Khatib SM, Almendral J, Aguinaga L, Berger RD, Cuesta A, Daubert JP, Dubner S, Ellenbogen KA, Estes NA 3rd, Fenelon G, Garcia FC, Gasparini M, Haines DE, Healey JS, Hurtwitz JL, Keegan R, Kolb C, Kuck KH, Marinskis G, Martinelli M, McGuire M, Molina LG, Okumura K, Proclemer A, Russo AM, Singh JP, Swerdlow CD, Teo WS, Uribe W, Viskin S, Wang CC, Zhang S. 2015 HRS/EHRA/APHRS/SOLAECE expert consensus statement on optimal implantable cardioverter-defibrillator programming and testing. J Arrhythm. 2016 Feb;32(1):1-28. doi: 10.1016/j.joa.2015.12.001. Epub 2016 Feb 1. No abstract available. PMID 26949427
- [Result] Sticherling C, Zabel M, Spencker S, Meyerfeldt U, Eckardt L, Behrens S, Niehaus M; ADRIA Investigators. Comparison of a novel, single-lead atrial sensing system with a dual-chamber implantable cardioverter-defibrillator system in patients without antibradycardia pacing indications: results of a randomized study. Circ Arrhythm Electrophysiol. 2011 Feb;4(1):56-63. doi: 10.1161/CIRCEP.110.958397. Epub 2010 Dec 14. PMID 21156772
- [Result] Healey JS, Connolly SJ, Gold MR, Israel CW, Van Gelder IC, Capucci A, Lau CP, Fain E, Yang S, Bailleul C, Morillo CA, Carlson M, Themeles E, Kaufman ES, Hohnloser SH; ASSERT Investigators. Subclinical atrial fibrillation and the risk of stroke. N Engl J Med. 2012 Jan 12;366(2):120-9. doi: 10.1056/NEJMoa1105575. PMID 22236222
- [Result] Miller DJ, Khan MA, Schultz LR, Simpson JR, Katramados AM, Russman AN, Mitsias PD. Outpatient cardiac telemetry detects a high rate of atrial fibrillation in cryptogenic stroke. J Neurol Sci. 2013 Jan 15;324(1-2):57-61. doi: 10.1016/j.jns.2012.10.001. Epub 2012 Oct 24. PMID 23102659
- [Result] Tayal AH, Tian M, Kelly KM, Jones SC, Wright DG, Singh D, Jarouse J, Brillman J, Murali S, Gupta R. Atrial fibrillation detected by mobile cardiac outpatient telemetry in cryptogenic TIA or stroke. Neurology. 2008 Nov 18;71(21):1696-701. doi: 10.1212/01.wnl.0000325059.86313.31. Epub 2008 Sep 24. PMID 18815386
- [Result] Ziegler PD, Rogers JD, Ferreira SW, Nichols AJ, Richards M, Koehler JL, Sarkar S. Long-term detection of atrial fibrillation with insertable cardiac monitors in a real-world cryptogenic stroke population. Int J Cardiol. 2017 Oct 1;244:175-179. doi: 10.1016/j.ijcard.2017.06.039. Epub 2017 Jun 10. PMID 28624331